CLINICAL TRIAL: NCT02752698
Title: Safety and Feasible Study of Domestic Surgical Robot That Had Been Authorized to Enter the Clinical Trial Stage
Brief Title: Domestic Surgical Robot Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: XY3-DSRCS1507A01
Record Dates: First submitted 2015-06-15; First posted 2016-04-27 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Gastric Ulcer With Perforation But Without Obstruction; Colon Cancer; Cholecystolithiasis; Appendicitis; Sleeve Gastrectomy; Gastric Bypass; Gastric Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Cholecystolithiasis; Appendicitis; Stomach Neoplasms; Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Micro Hand S robotic group (Experimental): Micro Hand S robotic surgery group
  Interventions: Procedure: Micro Hand S robotic surgery
- laparoscopic surgery (Other): laparoscopic surgery group
  Interventions: Procedure: laparoscopic surgery
- da Vinci robotic group (Other): da Vinci robotic robotic group
  Interventions: Procedure: da Vinci robotic surgery

INTERVENTIONS:
Procedure: Micro Hand S robotic surgery — 20-70 patients undergo Micro Hand S robotic surgeries
  Arms: Micro Hand S robotic group
Procedure: laparoscopic surgery — 20-70 patients undergo laparoscopic surgeries
  Arms: laparoscopic surgery
Procedure: da Vinci robotic surgery — 20-70 patients undergo da Vinci robotic surgeries
  Arms: da Vinci robotic group

SUMMARY:
Central South University in collaboration with Tianjin University developed the first domestically produced Chinese minimally invasive surgical (MIS) robot system which named "Micro Hand S" in 2013. Recently, as the domestic surgical robot research project's main section, this new MIS robot had been authorized to enter the clinical trial stage by the Ethics Committee of the Third Xiangya Hospital at Central South University.

DETAILED DESCRIPTION:
One surgeon perform these surgical trials using the robot "Micro Hand S". All of the patients were followed for 12 months, and pre- and postoperative changes in blood route test and hepatorenal function examination, surgery duration, hospital stay, total robotic setup time, total robotic operation time, intraoperative blood loss, total postoperative drainage amount, duration of bearing drainage tubes were recorded. In addition, the pre- and postoperative changes in the pathological and functional outcomes were measured.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of gastric tumor, colorectal tumor, acute cholecystitis and ileocecal tumor respectively
* 18years<age<65years
* male or female

Exclusion Criteria:

* patients with a history of open abdominal surgery
* unstable psychiatric illness
* an inability or reluctance to cooperate during long-term follow-up
* alcohol or drug addiction
* or relatively high surgical risks, such as abnormal coagulation function or bad heart, lung, liver and kidney function, were excluded from this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01-01; Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative outcomes | up to 1 week after operation
  surgical procedure/operative time/console time/blood loss/conversion
postoperative outcomes | up to 1 month after operation
  Time to first flatus/intake/hospital stay
pathological outcomes | up to 1 month after operation
  resection margin/harvested lymph node/mesorectal grade
complication | within 30 days after surgery
  type of complication/grade of complication

SECONDARY OUTCOMES:
functional outcomes | at least12 months after operation
  wexner/ipss/iief score
recurrence | at least 12 months after operation
  local recurrence and metastasis
survival | at least 12 months yesra after operation
  disease free survival/overall survival
change of blood and biochemiacl | within 1 month after operation
  wbc/hgb/albumin/cea

CONTACTS AND LOCATIONS:
Overall Officials: shaihong zhu, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lei Y, Jiang J, Zhu S, Yi B, Li J. Comparison of the short-term efficacy of two types of robotic total mesorectal excision for rectal cancer. Tech Coloproctol. 2022 Jan;26(1):19-28. doi: 10.1007/s10151-021-02546-0. Epub 2021 Nov 30. PMID 34846614
- [Derived] Zeng Y, Wang G, Li Z, Lin H, Zhu S, Yi B. The Micro Hand S vs. da Vinci Surgical Robot-Assisted Surgery on Total Mesorectal Excision: Short-Term Outcomes Using Propensity Score Matching Analysis. Front Surg. 2021 May 11;8:656270. doi: 10.3389/fsurg.2021.656270. eCollection 2021. PMID 34046424